CLINICAL TRIAL: NCT03266510
Title: Inspiratory Muscle Strength Training to Improve Blood Pressure and Physiological Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Douglas Seals (Other)
Responsible Party: Sponsor-Investigator, Douglas Seals, Professor of Distinction, University of Colorado, Boulder
Organization: University of Colorado, Boulder (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-0151
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Hypertension; Prehypertension; Aging
Keywords: Inspiratory muscle strength training
MeSH Terms: conditions — Hypertension; Prehypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory muscle strength training (Experimental): Using a handheld device, subjects were perform 30 breaths a day, six days a week. The device produces resistance that increases the effort of breathing in. The resistance to breathing will be strong.
  Interventions: Other: Inspiratory muscle strength training
- Sham training (Sham Comparator): Using a handheld device, subjects were perform 30 breaths a day, six days a week. The device produces resistance that increases the effort of breathing in. The resistance to breathing will be weak.
  Interventions: Other: Sham training

INTERVENTIONS:
Other: Inspiratory muscle strength training — Subjects will perform inspiratory muscle strength training for 6 weeks.
  Arms: Inspiratory muscle strength training
Other: Sham training — Subjects will perform sham training for 6 weeks.
  Arms: Sham training

SUMMARY:
The purpose of this study is to assess the efficacy of inspiratory muscle strength training for lowering blood pressure and improving physiological function (vascular, motor, and cognitive) in middle-aged and older adults with elevated systolic blood pressure.

DETAILED DESCRIPTION:
Over, the proposed research project has the long-term potential to influence clinical practice by establishing a novel lifestyle intervention for treating multiple domains of age- and hypertension-associated physiological dysfunction and thereby reducing the risk of clinical disease and disability.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Willing to accept random assignment to condition
* Women will be confirmed as postmenopausal (either natural or surgical) based on cessation of menses for >1 year.
* Resting systolic blood pressure 120-159 mmHg
* Resting diastolic blood pressure <100 mmHg
* Subjects taking anti-hypertensive medications will be included provided they meet the other inclusion criteria, including elevated systolic blood pressure. These medications will not be withheld prior to experimental protocols.
* Free from alcohol dependence or abuse, as defined by the American Psychiatry Association, Diagnostic and Statistical Manual or Mental Disorders (DSM-IV)

Exclusion Criteria:

* Current smoking
* Chronic clinical disease (e.g., inflammatory bowel disease/irritable bowel syndrome, coronary artery/peripheral artery/cerebrovascular diseases, diabetes, chronic kidney disease requiring dialysis, neurological disorders or diseases that may affect motor/cognitive function [multiple sclerosis, Parkinson's disease, polio, Alzheimer's disease, dementia, or other brain diseases of aging]), except hypertension
* Postmenopausal <1 year
* Scoring <21 on the mini-mental state examination
* Moderate or sever peripheral artery disease (ankle-brachial index 0.7)
* Taking a medication that your doctor deems unsafe to hold for >1 week
* A graded exercise test will be performed by all subjects. If there is physician concern or an adverse event, the subject will not participate in the study.
* No weight stable in the prior 3 months (>2 kg weight change) or unwilling to remain weight stable throughout study (rationale: recent weight change or weight loss can influence vascular function)

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2017-11-25 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 6 weeks
  Resting blood pressure

SECONDARY OUTCOMES:
Ambulatory blood pressure | 6 weeks
  24-hour mean blood pressure
Endothelium-dependent dilation | 6 weeks
  Flow-mediated dilation
Arterial stiffness | 6 weeks
  Aortic pulse wave velocity
Motor function | 6 weeks
  NIH Toolbox motor test battery
Cognitive function | 6 weeks
  NIH Toolbox cognition test battery
Systemic markers of oxidative stress | 6 weeks
  Oxidized LDL levels in blood
Endothelial cell markers of oxidative stress | 6 weeks
  Nitrotyrosine levels in biopsied endothelial cells

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H Craighead, PhD, Principal Investigator — University of Colorado, Boulder; Douglas R Seals, PhD, Study Director — University of Colorado, Boulder
Locations (1):
- Integrative Physiology of Aging Laboratory, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Craighead DH, Freeberg KA, Heinbockel TC, Rossman MJ, Jackman RA, McCarty NP, Jankowski LR, Nemkov T, Reisz JA, D'Alessandro A, Chonchol M, Bailey EF, Seals DR. Time-Efficient, High-Resistance Inspiratory Muscle Strength Training Increases Exercise Tolerance in Midlife and Older Adults. Med Sci Sports Exerc. 2024 Feb 1;56(2):266-276. doi: 10.1249/MSS.0000000000003291. Epub 2023 Sep 12. PMID 37707508
- [Derived] Craighead DH, Heinbockel TC, Freeberg KA, Rossman MJ, Jackman RA, Jankowski LR, Hamilton MN, Ziemba BP, Reisz JA, D'Alessandro A, Brewster LM, DeSouza CA, You Z, Chonchol M, Bailey EF, Seals DR. Time-Efficient Inspiratory Muscle Strength Training Lowers Blood Pressure and Improves Endothelial Function, NO Bioavailability, and Oxidative Stress in Midlife/Older Adults With Above-Normal Blood Pressure. J Am Heart Assoc. 2021 Jul 6;10(13):e020980. doi: 10.1161/JAHA.121.020980. Epub 2021 Jun 29. PMID 34184544
- See also: Description of our Research Laboratory — http://www.colorado.edu/intphys/research/cardiovascular.html